CLINICAL TRIAL: NCT05530252
Title: Effects of Antimicrobial Peptides Application After Non-surgical Periodontal Therapy on Treatment of Stage III and Grade B Periodontitis
Brief Title: Effects of AMP Application After Non-surgical Periodontal Therapy on Treatment of Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Stomatological Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Yongmei Xie, Principal Investigator, Beijing Stomatological Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUSH-IRB-KJ-PJ-2018-03
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patients did not know their group or the drugs they were given
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AMP Group (Experimental): scaling and root planning and subgingival application of antimicrobial peptide gel
  Interventions: Drug: Oral biological antimicrobial gel
- Perio Group (Active Comparator): scaling and root planning and subgingival application of minocycline hydrochloride ointment
  Interventions: Drug: minocycline hydrochloride ointment
- SRP Group (Other): scaling and root planning
  Interventions: Other: SRP

INTERVENTIONS:
Drug: Oral biological antimicrobial gel — The patients were divided into subgingival scaling, and Oral Biological Antimicrobial Gel was used in the periodontal pocket after scaling. The injection probe with gel was inserted into the periodontal pocket, and the injection was slowly pushed, and the injection was gradually withdrawn during the injection, until a little gel was found at the mouth of the bag.
  Other Names: Biokiller Oral Biological Antimicrobial Gel
  Arms: AMP Group
Drug: minocycline hydrochloride ointment — The patients were divided into subgingival scaling, and minocycline hydrochloride ointment was used in the periodontal pocket after scaling. The injection probe with gel was inserted into the periodontal pocket, and the injection was slowly pushed, and the injection was gradually withdrawn during the injection, until a little gel was found at the mouth of the bag.
  Other Names: Periocline
  Arms: Perio Group
Other: SRP — only scaling and root planning was performed on the patient
  Arms: SRP Group

SUMMARY:
Chronic periodontitis is an infectious disease of periodontal support tissues caused by bacterial biofilm, which leads to inflammation and destruction of periodontal support tissues ultimately resulting in tooth loss.In the clinic, patients with Stage III and Grade B periodontitis are difficult to gain desired outcomes on account of deep periodontal pockets, complicated anatomy, the removal of subgingival dental biofilms, and control of residual inflammation. A large number of studies have indicated that the effectiveness of local application of antibiotics as an adjunct to scaling and root planning (SRP), such as the antimicrobial and minocycline hydrochloride could affect bacterial metabolism and inhibit bioﬁlm attachment particularly in terms of pocket depth reduction and attachment level gain. However, the use of wide-spectrum antibiotics may cause some inevitable side effects including drug resistance, pathogens and probiotics were eliminated leading to diversity of microbiota diminished, and toothstaining. To solve the problems of antibiotics in the clinic, antimicrobial peptides (AMPs) may be considered as an alternative to conventional antibiotics drugs.In this randomized clinical trial, we aimed to evaluate the effects of AMPs as an addition to SRP on clinical parameters and microbiological biofilms in patients with Stage III and Grade B periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Previously untreated Stage III and Grade B periodontitis by clinically and radiologically。In 2018, EEP and AAP sorted out periodontitis into four classifications (Stage I to IV) based on several variables including clinical attachment loss, amount and percentage of bone loss, probing depth, presence and extent of angular bony defects and furcation involvement, tooth mobility, and tooth loss due to periodontitis, and three levels (grade A: low risk, grade B: moderate risk, grade C: high risk of progression) according to the rate of disease progression.
* A minimum of 20 natural teeth in the mouth, and more than 4 molars.

Exclusion Criteria:

* Acute oral lesions or necrotizing ulcerative periodontitis,
* Having received antibiotics within 6 months or the need for antibiotic coverage during experiment,
* Being allergic to minocycline,
* No orthodontic treatment,
* A history of systemic diseases,
* Pregnancy,
* Smoker

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- BeijingSHCMU, Beijing, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AMP Group | Perio Group | SRP Group
Started | 17 | 17 | 17
Completed | 16 | 16 | 16
Not Completed | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AMP Group | Perio Group | SRP Group | Total
Number analyzed (Participants) | 17 | 17 | 17 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.73 (14.03) | 37.93 (12.74) | 38.50 (10.01) | 38.39 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Because three subjects did not return to the clinic according to the time, they were not included in the final study analysis
  Participants
    Female | 11 | 10 | 10 | 31
    Male | 6 | 7 | 7 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Probing depth [Mean (Inter-Quartile Range); unit: millimeter] | 5.0 [5.0 to 5.1] | 4.9 [4.8 to 5.0] | 5.0 [4.9 to 5.1] | 5.0 [4.9 to 5.1]

OUTCOME MEASURES:

1. Primary Outcome: Periodontal Probing Depth
Description: from the gingival margin to the bottom of the periodontal pocket were assessed using a Williams periodontal probe((Hu-Friedy)
Time Frame: Change from Baseline Periodontal probing depth at 90 days
Population: Three subjects did not return to the clinic as required and were not included in the final data analysis of the study
Measure: Mean (Inter-Quartile Range); unit: millimeter
Arm/Group | AMP Group | Perio Group | SRP Group
Number analyzed (Participants) | 16 | 16 | 16
millimeter | 2.5 [2.4 to 2.6] | 3.2 [3.1 to 3.3] | 3.4 [3.3 to 3.4]

2. Primary Outcome: Attachment Level Were Assessed Using a Williams Periodontal Probe((Hu-Friedy)
Description: from the cementoenamel junction, crown margin or restoration to the bottom of the pocket
Time Frame: Change from Baseline Attachment level at 90 days
Population: Three subjects did not return to the clinic as required and were not included in the final data analysis of the study
Measure: Mean (Inter-Quartile Range); unit: millimeter
Arm/Group | AMP Group | Perio Group | SRP Group
Number analyzed (Participants) | 16 | 16 | 16
millimeter | 1.0 [0.9 to 1] | 1.7 [1.5 to 1.9] | 2.0 [1.7 to 2.2]

3. Primary Outcome: Bleeding Index Were Assessed Using a Williams Periodontal Probe((Hu-Friedy) ,the Rating Method Was Assessed Using the Criteria of Mazza.
Description: Bleeding index :
  0 = normal appearance of the gingiva and no bleeding on sulcus probing.
  1. = normal appearance of the gingiva but bleeding on probing of the sulcus.
  2. = bleeding on probing and gingival color change without swelling.
  3. = bleeding on probing, gingival color change with mild swelling.
  4. = bleeding on probing with marked gingival swelling, with or without color change.
  5. = bleeding on probing, L Spontaneous bleeding, gingival color change with marked swelling, with or without ulceration.
Time Frame: Change from Bleeding index at 90 days
Population: Three subjects did not return to the clinic as required and were not included in the final data analysis of the study
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | AMP Group | Perio Group | SRP Group
Number analyzed (Participants) | 16 | 16 | 16
score on a scale | 0.7 [0.6 to 0.9] | 1.1 [1.0 to 1.3] | 1.3 [1.2 to 1.4]

ADVERSE EVENTS:
Time Frame: 1 week ，3 months
Description: Severe drug allergy：Drug ulceration of the gums、the oral mucosa is red and swollen、laryngeal edema、local drug eruption
Arm/Group | AMP Group | Perio Group | SRP Group
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT05530252/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT05530252/ICF_001.pdf